CLINICAL TRIAL: NCT05130515
Title: An Open-Label, Single Arm, Phase II Trial of Niraparib in Combination With Anlotinib in Patients With Platinum-Resistant Recurrent or Platinum-Refractory Clear Cell Ovarian Cancer.
Brief Title: Anlotinib Combined With Niraparib Dual Therapy in Platinum-resistant Recurrent Ovarian Clear Cell Carcinoma.
Acronym: CC-ANNIE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Zai Lab (Shanghai) Co., Ltd. (Industry); Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-016
Record Dates: First submitted 2021-11-10; First posted 2021-11-23 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-11

CONDITIONS: Platinum-resistant Recurrent Clear Cell Ovarian Cancer
Keywords: clear cell ovarian cancer; Platinum-resistant cancer; Niraparib; Anlotinib
MeSH Terms: interventions — niraparib; anlotinib

STUDY DESIGN:
Intervention Model Description: Drug: Niraparib Niraparib 200mg po QD day1~21 Drug: Anlotinib Anlotinib 10mg po QD day1~14.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Niraparib 200mg po QD day1~21, Anlotinib 10mg po QD day1~14
  Interventions: Drug: Niraparib; Drug: Anlotinib

INTERVENTIONS:
Drug: Niraparib — Niraparib 200mg po QD, day1~21
Drug: Anlotinib — Anlotinib 10mg po QD, day1~14, 3 weeks/cycle

SUMMARY:
According to the definition of National Comprehensive Cancer Network (NCCN), ovarian clear cell carcinoma (OCCC) is a less common subtype of epithelial ovarian cancer (EOC) . The preliminary trial ANNIE (NCT04376073) shows a promising efficacy and safety profile for the ANNIE combo (anlotinib+niraparib). There is limited progress in targeted therapy for those less common ovarian cancers. In this study (CC-ANNIE), we aim to evaluate the antitumor activity and safety of niraparib combined with anlotinib in patients with platinum-resistant or platinum-refractory OCCC.

DETAILED DESCRIPTION:
The CC-ANNIE trial is a single-arm, single-center, exploratory phase II trial. Eligible patients (≥18 & ≤70 years) are histologically confirmed platinum-resistant recurrent OCCC and 20 subjects are planned to be enrolled. All subjects must have measurable lesions (according to Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) and are going to be treated with niraparib 200mg once daily, anlotinib 10mg on day 1-14 of each 21-day cycle thereafter until disease progression or intolerable toxicity. The primary endpoint is the objective response rate.

ELIGIBILITY:
Inclusion Criteria:

1. The patients understood the test process, signed the informed consent form and agreed to participate in the study.
2. 18 ~70 years old, female.
3. Histologically confirmed ovarian clear cell carcinoma.
4. The patients received platinum-based chemotherapy after primary debulking surgery, and experienced a recurrence or progression during the therapy; or experienced a recurrence or progression within 6 months after at least 4 cycles platinum-based therapy; or experienced a recurrence within 6 months after the end of the last platinum-based chemotherapy.

   Definition of recurrence or progression: clearly documented radiographic progression or carbohydrate antigen (CA125) increased continuously (confirmed after 1 week) and accompanied by clinical symptoms or physical examination, indicating disease progression.

   It is allowed to receive no more than 1 non-platinum regimen between 2 platinum-based regimens; Patients with disease recurrence or progression during platinum-based therapy or patients whose time from platinum-based treatment (at least 4 cycles) to disease recurrence and progression is less than 6 months are allowed to receive no more than 1 systematic treatment regimen.
5. Expected survival more than 16 weeks.
6. ECOG (Eastern Cooperative Oncology Group) physical status score 0-1.
7. Good organ function.

   * Neutrophil counts ≥1500/µL
   * Platelet counts ≥100,000/µL
   * Hemoglobin ≥10g/dl
   * Serum creatinine≤1.5 times of the upper limit value, or creatinine clearance rate ≥ 60ml/min (according to Cockcroft Gault formula)
   * Total bilirubin≤1.5 times of the upper limit value or direct bilirubin ≤1.0 times of the upper limit value
   * Aspartate transaminase and alanine transaminase≤ 2.5 times of the upper limit value, and ≤5 times of the upper limit value when liver metastasis exists
8. Pregnancy test results were negative and patients willing to use appropriate contraceptive methods while in the trial and within 3 months after the last administration of CC-ANNIE combo; or keep abstinence during the trial; or women with no potential fertility.
9. Ability to comply with protocol.
10. All of the adverse events caused by chemotherapy recovered to Common Terminology Criteria Adverse Events (CTCAE) grade 1 or baseline, except for stable sensory neuropathy or hair loss ≤ CTCAE grade 2.
11. At least 1 measurable lesions (according to RECIST 1.1)
12. The interval between initial administration of CC-ANNIE combo and previous chemotherapy, radiotherapy, targeted therapy, immunotherapy, or other antitumor therapy should be at least 4 weeks, or at least 6 weeks if the chemotherapy regimen includes mitomycin.

Exclusion Criteria:

1. Any poly(adenosine diphosphate-ribose) polymerase (PARP) inhibitors treatment history.
2. Allergy to active or inactive ingredients of niraparib or drugs with similar chemical structures.
3. Allergy to active or inactive ingredients of anlotinib or drugs with similar chemical structures.
4. Active and uncontrollable brain metastasis or leptomeningeal metastasis. Patients with spinal cord compression can still be considered if they have received targeted treatment and have evidence of clinical stability of the disease for at least > 28 days (controlled brain metastasis must have received radiotherapy or chemotherapy at least 1 month prior to study entry; patients may not have new symptoms related to brain lesions or symptoms indicating disease progression and either take a stable dose of hormone or do not need to take hormone).
5. Major surgery performed within 3 weeks before enrollment, or any surgical effects that have not been recovered from the surgery, or chemotherapy.
6. >20% bone marrow palliative radiotherapy performed within 1 week before enrollment.
7. Any other malignant tumor exclude ovarian cancer has been diagnosed within 2 years before enrollment (except for completely treated basal or squamous cell skin cancer).
8. Combined with central squamous cell carcinoma of lungs or at risk of massive hemoptysis (such as bronchiectasis and uncured tuberculosis).
9. Myelodysplastic syndromes (MDS) or acute myelocytic leukemia (AML).
10. Serious or uncontrollable diseases, including but not limited to:

    * uncontrollable nausea and vomiting, inability to swallow the study drug, any gastrointestinal disease that may interfere with drug absorption and metabolism.
    * active viral infections such as human immunodeficiency virus, hepatitis B, hepatitis C, etc.
    * uncontrolled major seizures, unstable spinal cord compression, superior vena cava syndrome or other mental disorders that affect the patient's informed consent.
    * immune deficiency (except splenectomy), or other diseases that researchers believe may expose patients to high-risk toxicity.
11. Prone to bleeding and history of thrombosis:

    * Any CTCAE grade 2 bleeding events occurred within 3 months, or ≥ CTCAE grade 3 bleeding events occurred within 6 months.
    * A history of gastrointestinal bleeding or a clear tendency of gastrointestinal bleeding within 6 months. For example, esophageal varices with bleeding risk, local active ulcer lesions, or occult blood in stool++
    * Active bleeding or abnormal coagulation function, have bleeding tendency, or are receiving thrombolytic or anticoagulant therapy
    * Need anticoagulant therapy with warfarin or heparin
    * Need long-term antiplatelet therapy (such as aspirin and clopidogrel)
    * Thrombotic or embolic events occurred in the past 6 months, such as cerebrovascular accidents (including transient ischemic attack) and pulmonary embolism.
12. History of severe cardiovascular disease:

    * New York Heart Association (NYHA) Grade 3 and 4 congestive heart failure.
    * Unstable angina or newly diagnosed angina or myocardial infarction within 12 months prior to study.
    * Arrhythmias requiring therapeutic intervention (patients taking beta-blockers or digoxin can be included).
    * CTCAE≥2 valvular heart disease.
    * Poorly controlled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg).
13. Abnormal laboratory tests:

    * Hyponatremia (sodium < 130 mmol/L); Baseline serum potassium < 3.5mmol /L (potassium supplement can be used before entering the study).
    * Abnormal thyroid function that cannot be maintained within normal limits with medication.
14. Any prior or current disease, treatment, or laboratory abnormality that may interfere with the study results or affect the patient's full participation in the study, or that the investigator deems the patient unsuitable for the study. Patients should not receive platelet or red blood cell transfusions within 4 weeks before the start of treatment with the study drug.
15. Pregnancy or lactation, or expected pregnancy during study treatment.
16. Q-T interval corrected (QTc)>450 ms. If the patient has prolonged QTc interval, but the investigator assessed the reason for the prolonged period as pacemaker (without other cardiac abnormalities), discussion with the investigator will be required to determine whether the patient is suitable for study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate | at 6 months
  The primary objective of this study is to determine the preliminary efficacy of administration of niraparib in combination with anlotinib in the treatment of platinum-resistant recurrent or platinum-refractory clear cell ovarian cancer, as measured by the objective response rate (ORR), which is a combination of CR (complete response, the target lesion completely disappeared over 4 weeks) and PR (partial response, the target lesions were reduced by more than 30% for more than 4 weeks).

SECONDARY OUTCOMES:
The frequency and severity of adverse events | Baseline through 1.5 year
  The frequency and severity of adverse events and toxicity based upon CTCAE version 5.0 during subjects receiving the study treatment.
Duration of response | at 12 months
  Duration of response is defined as the time from the first documentation of CR or PR to the first documentation of tumor progression, or to death due to any cause.
Time to response | at 6 months
  Time to response is defined as the time from date of enrollment to the date of first documented tumor response (CR or PR).
24 weeks clinical benefit rate | at 24 weeks
  24 weeks clinical benefit rate is defined as the rate of CR plus PR and stabel disease (SD).
Objective response rate of homologous recombination deficient group | at 6 months
  The efficacy of administration of niraparib in combination with anlotinib in the homologous recombination deficient group.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the medresman site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available, within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://www.medresman.org.cn